CLINICAL TRIAL: NCT03674788
Title: The Prospective LEUVEN Transcatheter Valve Therapy Registry
Acronym: LEUVEN-TVT
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S61523
Record Dates: First submitted 2018-07-17; First posted 2018-09-18 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- TAVI: Transcatheter Aortic Valve Implantation
  Interventions: Device: Transcatheter valve intervention
- TMVI: Transcatheter Mitral Valve Intervention
  Interventions: Device: Transcatheter valve intervention
- TTVI: Transcatheter Tricuspid Valve Intervention
  Interventions: Device: Transcatheter valve intervention

INTERVENTIONS:
Device: Transcatheter valve intervention

SUMMARY:
Assessment of feasibility, safety and outcomes of transcatheter valve interventions

DETAILED DESCRIPTION:
Transcatheter valve therapies have a growing impact on daily medical practice since the first human percutaneous implantation of an aortic valve bioprosthesis by A. Cribier in 2002. While initially these techniques were reserved for patients at prohibitive risk for surgical aortic valve implantation, indications moving toward patients at high and intermediate risk.

Outcomes of these percutaneous interventions need to be monitored to assess quality of care and tailor indications in this rapidly moving field in interventional cardiology.

Trial objectives and Design Trial objectives

* to describe patient populations selected for transcatheter valve treatment
* to describe procedural aspects and results
* to perform clinical and hemodynamic follow-up of the patients Primary endpoints The primary endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium criteria (2-3).

Secondary endpoints The secondary endpoints of the study are hemodynamic outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium criteria (2-3). Quality of life parameters, as well as exercise tolerance will be assessed.

Trial Design The design of the trial is a prospective non-interventional registry.

ELIGIBILITY:
Inclusion Criteria:

* All patients selected for percutaneous treatment of a valve disorder potentially qualify for the present registry

Exclusion Criteria:

* All patients selected for percutaneous treatment of a valve disorder potentially qualify for the present registry. There are no formal exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing transcatheter valve intervention
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2008-03-12 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 10 years of follow-up
  The primary endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Cardiovascular death | 10 years of follow-up
  The primary endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
All-cause death and/or rehospitalisation for cardiovascular causes | 10 years of follow-up
  The primary endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
All-cause death and/or major stroke | 10 years of follow-up
  The primary endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).

SECONDARY OUTCOMES:
Rehospitalisation for cardiovascular causes | 10 years of follow-up
  The endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Stroke | 10 years of follow-up
  The endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Kidney injury | early after index intervention (30 days)
  AKIN classification. The endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Bleeding complications | early after index intervention (30 days)
  BARC classification. The endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Vascular complications | early after index intervention (30 days)
  The endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Myocardial infarction | early after index intervention (30 days)
  The endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Conduction disturbances and arrhythmias | early after index intervention (30 days)
  The endpoints of the study are clinical outcomes after transcatheter valve interventions according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Quality of life | 10 years of follow-up
  EQ5D and EQ-Visual analogue scale
Exercise tolerance | 2 years of follow-up
  6-minutes walking test
Valvular function according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18). | 10 years of follow-up
  Mean and peak gradient (mmHg) Effective orifice area (cm²) Left ventricular ejection fraction (%) valvular regurgtiation
Device success | 30 days of follow-up
  Combined endpoint according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Early safety | 30 days of follow-up
  Combined endpoint according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Clinical efficacy | 10 years of follow-up
  Combined endpoint according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).
Time-related valve safety | 10 years of follow-up
  Combined endpoint according to the Valve Academic Research Consortium 2 criteria (Eur Heart J. 2012 Oct;33(19):2403-18).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, University Hospital Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No